CLINICAL TRIAL: NCT05658601
Title: SWITCH - ITA A Multicentre, Single Country, Prospective Non Interventional Observational Study to Describe the Switching From a First- or Second-line Disease Modifying Therapy (DMT) to Ozanimod, in Relapsing Remitting Multiple Sclerosis (RRMS) Patients Treated According to Clinical Practice.
Brief Title: A Study to Describe the Switching From a First- or Second-line Disease Modifying Therapy (DMT) to Ozanimod in Participants With Relapsing Remitting Multiple Sclerosis (RRMS)
Acronym: SWITCH - ITA
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-1038
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Ozanimod
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1

SUMMARY:
The purpose of this study is to describe the reasons, therapy, and/or disease for changing first or second line Disease Modifying Therapy (DMT) to ozanimod in participants with Relapsing Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with RRMS according to 2017 revised McDonald criteria
* Patients who switched a previous first or second line DMT to ozanimod between 4 and 12 weeks before the enrollment
* Patient with a MRI performed within three months before the enrollment
* Patient eligible to ozanimod according to SmPC

Exclusion Criteria:

* Patients with clinical forms of MS other than RRMS
* Patients unable to participate for various reasons
* Patients participating in another clinical study with an investigational product if the study considers the switching behavior as an endpoint or objective
* Contraindications to ozanimod according to SmPC

Other protocol-defined Inclusion/Exclusion Criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is composed of 180 participants 18-55 years with Relapsing Remitting Multiple Sclerosis (RRMS) diagnosed according to 2017 revised McDonald criteria, switching from a first or second line Disease Modifying Therapy (DMT) to ozanimod, and in treatment with ozanimod between 4 and 12 weeks before the enrollment.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Reason for switching treatment | At baseline
  Reason for switching the previous treatment: Lack of efficacy, Poor safety/tolerability, Difficulty in administration, Poor compliance, Patient's request, or other reasons
Mode of switching treatment | At baseline
  Wash-out from previous treatment (first/second line DMT) (days), overlapping (days), dosage (first/second line DMT and ozanimod), concomitant treatments

SECONDARY OUTCOMES:
Expanded Disability Status Score (EDSS) | At baseline, week 12, and week 24
  Mean EDSS score in patients enrolled in the study
MRI | At baseline, week 12, and week 24
  Number of new or enlarging T2 lesions and T1 Gadolinium Enhancing Lesions (GdE) lesions.
TSQM | At baseline and week 24
  Treatment Satisfaction Questionnaire for Medication
Lymphocyte sub populations | At baseline, week 12, and week 24
  The pattern of the sub populations of lymphocytes: CD3, CD4, CD8, CD19, CD56.
Incidence of Adverse Events (AEs) | Continuous (Up to 42 months)
  Number of AEs in the study population during the study; AEs will be coded according to MEdDRA.
Incidence of Serious Adverse Events (SAEs) | Continuous (Up to 42 months)
  Number of SAEs in the study population during the study; SAEs will be coded according to MEdDRA.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Isernia, Italy

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html